CLINICAL TRIAL: NCT03844971
Title: Evaluation of Accuracy of Computer Guided Arthrocentesis of Temporomandibular Joint for Patients With Anterior Disc Displacement With Reduction Using Patient Specific Guide (Case Series)
Brief Title: Computer Guided Arthrocentesis of Temporomandibular
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mahmoud, Resident, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-02-16
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Temporomandibular Disorder
Keywords: Arthrocentesis; Computer assisted surgery; Anterior disc displacement with reduction
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: Case series A trial will be carried out in hospital of oral and maxillofacial surgery department faculty of dentistry
Masking Description: Single grouped study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer assisted surgery (Experimental): Intervention will be fabrication of patient specific surgical guide for arthrocentesis of temporomandibular joint for patients with anterior disc displacement with reduction using patient computed tomography with the aid of computer aided surgical simulation software
  Interventions: Procedure: Computer assisted arthrocentesis of

INTERVENTIONS:
Procedure: Computer assisted arthrocentesis of — Under general anesthesia : patients specific preoperative prefabricated surgical guide will be used intraoperative for arthrocentesis of temporomandibular joint for patients with anterior disc displacement with reduction
  Other Names: Computer guided surgery

SUMMARY:
Computer guided arthrocentesis of temporomandibular joint for patients with anterior disc displacement with reduction using patient specific guide

DETAILED DESCRIPTION:
A consecutive, single centered prospective study. All the patients will be selected from the Outpatient Clinic of the Oral and Maxillofacial Surgery Department. Faculty of dentistry- Cairo University Egypt.

Patients will be subjected to:

* Case history including personal data, medical, surgical and family history.
* Clinical examination
* Radiographic examination using magnetic resonance imaging (MRI) and computed tomography (C.T) bony and soft tissue window.
* Diagnostic studying casts, laser scanning of the casts in centric occlusion
* Preoperative anaesthesia assessment for fitness for general anaesthesia.
* Utilizing computer aided surgical simulation software a patient specific surgical guide is designed from the patients' segmented 3D soft tissue window with the following criteria:
* and fabrication of the surgical guide using c.t. scan with soft tissue and bony window, segmentation of the 3D model using Mimics 19.0 (medical engineering program), designing a 3D patient specific the guide is resting on skin of buccal and temporal area and occlusal bite block with a 3 openings i. The guide is resting on skin of buccal and temporal area and occlusal bite block with 3 openings ii. 2 depth controlled cylinders for input and output needles iii. 1 cylinder for arthroscopy trocar arm for verification of needle tip location in the superior joint space
* Then exporting the stl file to 3D printing machine before surgery All cases will undergo surgery under general anesthesia. The patient specific guide will be adapted on facial soft tissue overlying the temporomandibular joint . Fixation of the guide using occlusal bite-block on maxillary and mandibular teeth. Insertion of arthroscopic trocar through the depth controlled cylinder. Locating the superior joint space using arthroscopy. Insertion of input needle through the depth controlled cylinder. Verification of the needle position and angulation in the superior joint space by the arthroscopy. Infusion of 2ml lactated Ringer's solution then insertion of output needle and joint effusion by 300 ml of lactated Ringer's solution then infusing the joint by 2ml of hyaluronic acid.

Proper postoperative instructions will be given to the patient as soft diet for 1 week and immediate postoperative physiotherapy from the second day of operation and for 1 month. in addition to the postoperative medications including antibiotics (amoxicillin 500mg capsules t.i.d) and analgesics (diclofenac potassium 50mg as needed).Adherence to follow ups is also instructed

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior disc displacement with reduction
* Age group : from 15 to 60 years old
* No sex predilection
* Patients with no contraindications to surgical intervention

Exclusion Criteria:

* Patients with systemic condition counteracting with the surgical procedure.
* Patients with disc displacement without reduction
* Patients with osteoarthritis
* Patients suffering from myofacial pain
* Pregnant or lactating female

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-03-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Intraoperative
  The primary outcome is the accuracy of the needle position in the superior joint space. It is binary outcome measured as yes or no. Aggregation will be done by percentage of successful cases number in the study. Calculation of the mean of all cases will be performed for analysis of the results
Patient satisfaction | 6 months postoperatively
  Recording preoperative and 9 consecutive postoperative numerical records over 6 months will be done. Percentage of successful cases number in the study will be aggregated. Calculation of the mean of all cases will be performed for analysis of the results.

SECONDARY OUTCOMES:
Maximal mouth opening | 6 month postoperatively
  Measuring preoperative and 9 consecutive postoperative maximal mouth opening over 6 months will be done. The measuring unit is millimetres. Percentage of successful cases number in the study will be aggregated. Calculation of the mean of all cases will be performed for analysis of the results.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Mounir, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Giza, ElManial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bas B, Kazan D, Kutuk N, Gurbanov V. The Effect of Exercise on Range of Movement and Pain After Temporomandibular Joint Arthrocentesis. J Oral Maxillofac Surg. 2018 Jun;76(6):1181-1186. doi: 10.1016/j.joms.2018.01.003. Epub 2018 Jan 12. PMID 29406255
- [Background] Beumer HW, Puscas L. Computer modeling and navigation in maxillofacial surgery. Curr Opin Otolaryngol Head Neck Surg. 2009 Aug;17(4):270-3. doi: 10.1097/MOO.0b013e32832cba7d. PMID 19444109
- [Background] Chang CL, Wang DH, Yang MC, Hsu WE, Hsu ML. Functional disorders of the temporomandibular joints: Internal derangement of the temporomandibular joint. Kaohsiung J Med Sci. 2018 Apr;34(4):223-230. doi: 10.1016/j.kjms.2018.01.004. Epub 2018 Feb 7. PMID 29655411
- [Background] De Barros Melo MN, Dos Santos Melo JN, Sarmento VA, De Azevedo RA, Queiroz CS. Influence of arthrocentesis irrigation volume at temporomandibular disorder treatment. Indian J Dent Res. 2017 Nov-Dec;28(6):655-660. doi: 10.4103/ijdr.IJDR_422_15. PMID 29256465
- [Background] Efeoglu C, Calis AS, Koca H, Yuksel E. A stepped approach for the management of symptomatic internal derangement of the temporomandibular joint. J Otolaryngol Head Neck Surg. 2018 May 15;47(1):33. doi: 10.1186/s40463-018-0282-y. PMID 29764480
- [Background] Folle FS, Poluha RL, Setogutti ET, Grossmann E. Double puncture versus single puncture arthrocentesis for the management of unilateral temporomandibular joint disc displacement without reduction: A randomized controlled trial. J Craniomaxillofac Surg. 2018 Dec;46(12):2003-2007. doi: 10.1016/j.jcms.2018.10.015. Epub 2018 Oct 26. PMID 30446325